CLINICAL TRIAL: NCT01822145
Title: PREDICTion of Implantable-Cardioverter Defibrillator Shock Study
Brief Title: A Feasibility Study on Prediction of an ICD Shock by ICD-derived Data
Acronym: PREDICT-ICDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ngai Yin Chan, Principal investigator, Princess Margaret Hospital, Hong Kong
Other Study IDs: PREDICTICDS01
Record Dates: First submitted 2013-03-24; First posted 2013-04-02 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Sudden Cardiac Arrest; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: implantable-cardioverter-defibrillator; ventricular tachycardia; ventricular fibrillation; sudden cardiac arrest
MeSH Terms: conditions — Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD recipients: ICD recipients with documented cardiac arrest or ventricular arrhythmias
  Interventions: Device: ICD

INTERVENTIONS:
Device: ICD

SUMMARY:
The primary hypothesis is that an ICD shock may be predicted days in advance by a combined score derived from different data obtainable from the ICD

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧ 18 and ≦ 80
2. Patients have documented spontaneous and sustained ventricular arrhythmias in the last six months prior to the enrollment
3. Patients who are in sinus rhythm, have dual-chamber ICD or CRT-D implanted at least one month before enrollment
4. Patients who are in atrial fibrillation, have single-chamber ICD or CRT-D implanted at least one month before enrollment
5. Patients who are compliant to CareLink follow-up

Exclusion Criteria:

1. Patients who are pregnant
2. Patients who are incapable of giving consent to the study
3. Patients who have a life-expectancy of less than 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD recipients with documented cardiac arrest, ventricular tachycardia or ventricular fibrillation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
ICD-derived T-wave alternans amplitude before ICD shock | 6 months
  The T-wave alternans amplitude before an ICD shock will be measured in mV and compared to the baseline T-wave alternans amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Ngai Yin Chan, MBBS, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Hong Kong, China